CLINICAL TRIAL: NCT04163211
Title: Abdominal Drainage During Appendicectomy - Resources Down the Drain: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Principal Investigator, Scarlet Nazarian, Principal Investigator, The Whittington Hospital NHS Trust
Other Study IDs: 12345678
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Group 1: Patients with complicated appendicitis who had a drain inserted
  Interventions: Procedure: Abdominal drain
- Group 2: Patients with complicated appendicitis who did not have a drain inserted
  Interventions: Procedure: Abdominal drain

INTERVENTIONS:
Procedure: Abdominal drain — A latex-free drain (size 20F)

SUMMARY:
The investigators performed a retrospective review of all patients undergoing appendicectomy from March-November 2018 using the online theatre database and discharge letters. CA was defined as patients with perforated or gangrenous appendicitis on histology. Patients were divided into 2 groups; Group 1 (G1) included patients with CA who had a drain inserted; Group 2 (G2) included patients with CA and no drain.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 16 with complicated appendicitis (CA) were included

Exclusion Criteria:

* Patients with evidence of caecal/ appendicular malignancy were excluded.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients over the age of 16 with complicated appendicitis (CA) were included. CA was defined as histologically proven gangrenous or perforated appendicitis.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal abscess | Up to 6 months post-operative

SECONDARY OUTCOMES:
Length of stay | 8 months - March to November 2018
  Number of days patient in hospital since admission

CONTACTS AND LOCATIONS:
Locations (1):
- Whittington Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data if appropriate with permission of the Trust